CLINICAL TRIAL: NCT03735862
Title: Complications and 1-Year Outcomes Following Hiatal Hernia Repair With MIROMESH a Novel, Highly Vascular, Porcine Derived, Biologic Matrix
Brief Title: Complications, Outcomes and Revisions Following Hiatal Hernia Repair With MIROMESH
Status: Completed | Type: Observational
Sponsor: Miromatrix Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20174001
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Hiatal Hernia With Gastroesophageal Reflux Disease; Gastroesophageal Reflux; GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observations Group: Patients who have undergone a hiatal hernia repair with MIROMESH.
  Interventions: Biological: Hepatic derived surgical matrix

INTERVENTIONS:
Biological: Hepatic derived surgical matrix — Hiatal hernia repair with MIROMESH
  Other Names: MIROMESH Biologic Matrix

SUMMARY:
Investigator will identify a consecutive cohort of patients who have undergone a hiatal hernia repair and are at least 6 months post index procedure.

DETAILED DESCRIPTION:
Planned Sample Size: At minimum of 70 consecutive subjects at least 6-months post-index procedure

Study Population: A consecutive cohort of patients who have undergone a hiatal hernia repair with MIROMESH.

Primary Objective: Characterize the procedural and early post-operative safety profile of MIROMESH when used as reinforcement in hiatal hernia repair.

Secondary Objectives

A retrospective chart review will identify the appropriate cohort with a prospective follow-up survey to acquire safety and outcome information.

A retrospective chart review of appropriate subjects.

Data to be acquired will be:

Preoperative - Chart Review

* Gender
* Date of birth
* Weight
* Body Mass Index
* Specific diagnosis
* DeMeester Score
* 24 hour pH test (% acid exposure in 24 hours)
* Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) Score Peri-operative Preoperative - Chart Review
* Date of surgery
* Number of stitches used to close wound
* Paraesophageal hernia type
* Mesh shape
* Mesh size used
* Attachment technique
* Length of stay
* Complications

Post-Operative (With-in 1 month of surgery) Preoperative - Chart Review

* Complications (Mesh related)
* Complications (procedure related)
* Prolonged dysphagia (Y/N)
* Stenosis (Y/N)
* Dilations (Y/N)
* Esophagogastroduodenoscopy or Upper gastrointestinal series documented hernia recurrence
* GERD-HRQL Score

Prospective institutional review board approved Follow-Up Telephone Interview

* Have you had a revision surgery?
* GERD-HRQL Score
* How satisfied are you with the procedure?
* Have you used proton pump inhibitors in the last 3 months
* How likely are you to recommend this procedure to a loved one?

ELIGIBILITY:
Inclusion Criteria:

* Had a hiatal hernia repair with MIROMESH greater than 6 months prior to study

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Had a hiatal hernia repair with MIROMESH greater than 6 months prior to study
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George K Gillian, M.D., Principal Investigator — Virginia Heartburn and Hernia Institute
Locations (1):
- Virginia Heartburn and Hernia Institute, Lorton, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A consecutive cohort of patients who underwent a hiatal hernia repair between 1 Nov 2015 and 1 Mar 2017 at the principle investigator's private practice were identified. Patients were contacted by phone and asked if they were willing to participate. If so they were consented and enrolled.
Pre-assignment Details: 12 patients declined participation or could not be contacted. These were included in the baseline analysis.
Period: Overall Study
Arm/Group | Observations Group
Started | 73
Completed | 73
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 85 patients were identified - 73 agreed to participate and enrolled, the entire cohort was analyzed at baseline.
Arm/Group | Observations Group
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 85
GERD-HRQL [Mean (Standard Deviation); unit: Score] — Measure Description: The Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) scale assess on symptoms associated with gastroesophageal reflux disease. There are 10 questions (each representing a GERD symptom such as heartburn) answered on a 6-point scale of 0 - 6 with 0 indicating no symptoms and 5 indicating incapacitating symptoms. The answer to all questions are summed to give you a final score on the scale. Scores may range for 0 (no symptoms) to 50 (incapacitating symptoms).
  Score | 27.7 (9.3)
Proton Pump Inhibitor Use [Count of Participants; unit: Participants]
  Yes | 73
  No | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Required a Revision of the Index Surgery.
Description: Patient self-report if they had a revision or other laparoscopic surgery following index procedure.
Time Frame: 6-18 months post index procedure
Population: 12 patients declined participation or could not be contacted.
Measure: Count of Participants; unit: Participants
Arm/Group | Observations Group
Number analyzed (Participants) | 73
Participants | 0

2. Secondary Outcome: Gastroesophageal Reflux Disease Health Related Quality of Life Score (GERD-HRQL)
Description: The GERD-HRQL score assess the severity of GERD symptomatic and impact on the subjects quality of life. The score is comprised of 10 questions whose answers are summed for the final score. THe score can range from 0 to 50, with 50 being the worst and 0 meaning no impact.
Time Frame: 6-18 months post index procedure
Population: 12 patients declined participation or could not be contacted.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Observations Group
Number analyzed (Participants) | 73
Score | 7.1 (8.1)
Statistical Analysis 1: Comparison: Observations Group; Difference between baseline and follow-up; Test type: Other — Paired t-Test; p < 0.001, t-test, 1 sided

3. Secondary Outcome: Medication Use
Description: Use of PPIs in 3-months prior to follow-up interview
Time Frame: 6-18 months post index procedure
Population: 12 patients declined participation or could not be contacted. One patient did not answer.
Measure: Count of Participants; unit: Participants
Arm/Group | Observations Group
Number analyzed (Participants) | 72
Participants
  Yes | 7
  No | 65
Statistical Analysis 1: Comparison: Observations Group; Difference between baseline and follow-up; Test type: Superiority; p < 0.0001, McNemar

4. Other Pre Specified Outcome: Satisfaction With Procedure
Description: Patients reported their satisfaction with the procedure as "Dissatisfied", "Neutral", or Satisfied.
Time Frame: 6-18 Months post index procedure
Population: 12 patients declined participation or could not be contacted.
Measure: Count of Participants; unit: Participants
Arm/Group | Observations Group
Number analyzed (Participants) | 73
Participants
  Satisfied | 63
  Neutral | 6
  Dissatisfied | 4

5. Other Pre Specified Outcome: Likelihood to Recommend
Description: Patients were asked to report how likely they would be to recommend this procedure to a friend or loved one with the same condition. Report was based on a scale of 1 (not at all likely) to 10 (very likely).
Time Frame: 6-18 Months post index procedure
Population: 12 patients declined participation or could not be contacted.
Measure: Count of Participants; unit: Participants
Arm/Group | Observations Group
Number analyzed (Participants) | 73
Participants
  <=3 | 3
  >= 4 - <= 7 | 6
  >=8 | 64

ADVERSE EVENTS:
Time Frame: Operative & Peri-Operative, from admission for the surgical event through discharge. (Median length of stay 1 day)
Arm/Group | Observations Group
All-Cause Mortality (participants affected / at risk) | 0/73
Serious Adverse Events (participants affected / at risk) | 0/73
Other Adverse Events (participants affected / at risk) | 3/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observations Group (N=73)
Liver lobe tear (Surgical and medical procedures) | 1 (1)
Minor bleeding gastric vessels (Surgical and medical procedures) | 1 (1)
Arterial flutter (Surgical and medical procedures) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a retrospectively identified cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT03735862/Prot_SAP_000.pdf